CLINICAL TRIAL: NCT06539208
Title: A Phase I/IIa，Open-label, Single Ascending Dose and Dose-expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of YOLT-201 in Patients With Transthyretin Amyloidosis Polyneuropathy (ATTR-PN) or Transthyretin Amyloidosis Cardiomyopathy (ATTR-CM)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: YolTech Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YT-YOLT-201-101
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Transthyretin Amyloidosis Polyneuropathy; Transthyrexin Amyloidosis Cardiomyopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YOLT-201 (Experimental)
  Interventions: Drug: YOLT-201

INTERVENTIONS:
Drug: YOLT-201 — Infusion of YOLT-201 at Day 1

SUMMARY:
This study will be conducted to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of YOLT-201 in participants with hereditary transthyretin amyloidosis with polyneuropathy (ATTRv-PN) and participants with hereditary transthyretin amyloidosis with cardiomyopathy (ATTRv-CM).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 80 years old (including the critical values), regardless of gender;
2. Body weight at the time of screening is between 40 - 90kg (including the critical values);
3. TTR gene mutation is confirmed by genetic testing;
4. At the time of screening, the following laboratory standards must be met:

   1. AST, ALT, and TBIL ≤ the upper limit of the normal value (ULN);
   2. For subjects with Gilbert syndrome, TBIL ≤ 2 times ULN;
   3. Glomerular filtration rate (GFR) ≥ 45 mL/min/1.73m2 (calculated according to the CKD-EPI formula);
   4. Platelet count ≥ 100 × 109/L;
   5. Partial thromboplastin time (APTT), prothrombin time (PT), and thrombin generation time (TGT) are all within the reference value range, fibrinogen (FIB) ≥ the lower limit of the normal value (LLN) and ≤ 1.5*ULN, the international normalized ratio (INR) ≤ ULN, and if taking anticoagulant drugs, it is ≤ 2.5*ULN;
   6. Vitamin A and vitamin B12 ≥ the lower limit of the reference value (LLN);
   7. Low-density lipoprotein cholesterol (LDL) < 200 mg/dL (5.17 mmol/L).
5. Drugs approved for the treatment of ATTR are not accessible (Criterion A) and/or the disease still progresses despite the use of drugs approved for the treatment of ATTR (Criterion B):

   * Criterion A: Meeting one or more of the following criteria:

     1. Drugs for the treatment of ATTR are not marketed in China;
     2. Unable to receive the approved drugs for ATTR treatment (e.g., intolerance or other medical, cost and/or other reasons);
   * Criterion B: Subjects have received ATTR drug treatment for at least 3 months, but the subject's condition has progressed as assessed by the investigator, and meets any of the following criteria:

   ATTR-CM: a. Increased number of hospitalizations related to heart failure; b. Worsening of NYHA classification; c. Decrease in KCCQ score by at least 5 points; d. Decrease in 6-MWT by at least 30m; e. Increase in NT-proBNP by 30%; f. Increase in Troponin I by 30%; g. Echocardiography indicates an increase in left ventricular wall thickness by 2mm; h. Echocardiography indicates a decrease in left ventricular ejection fraction by ≥ 5% or a decrease in global longitudinal strain by ≥ 1% or a decrease in stroke volume by ≥ 5%; i. New conduction block appears; ATTR-PN: a. PND score increase by ≥ 1 point; b. FAP increases by 1 stage; c. NIS score increase by ≥ 5 points; d. NIS-Lower Limb score increase by ≥ 5 points; e. mBMI decrease by ≥ 25 kg/m2×g/L; f. 10-MWT decrease by ≥ 0.1 m/s; g. Electroneurophysiological examination (electromyography) worsens compared to the previous.
6. Agree to stop drinking alcohol within the screening period to 28 days after administration;
7. Female subjects need to be menopausal (absence of menstruation for at least 1 year) or have undergone uterine/ovarian resection surgery; Male subjects and their partners have no fertility plans from the screening period to 6 months after the end of the trial and agree to take effective non-pharmaceutical contraceptive measures during the trial;
8. The subject himself/herself (or his/her legally recognized representative) understands and signs the informed consent form;
9. Agree not to receive other ATTR drug intervention treatment within at least 8 weeks after administration of YOLT-201;

   For ATTR-PN only:
10. Diagnosed as ATTR-PN according to the "Consensus on the Diagnosis and Treatment of Transthyretin Amyloidosis Polyneuropathy", and the NIS score at the screening is ≥ 5 and ≤ 130, and the PND score is ≤ IIIb;
11. NT-proBNP < 600pg/ml at the screening;

    For ATTR-CM only:
12. Diagnosed as ATTR-CM according to the "Expert Consensus on the Diagnosis and Treatment of Transthyretin Cardiac Amyloidosis";
13. The New York Heart Association (NYHA) cardiac function classification is grade II - III;
14. The 6-minute walk test (6-MWT) is ≥ 150 m at the screening;
15. NT-proBNP is ≥ 600pg/mL and ≤ 3000pg/mL at the screening;
16. At the screening, echocardiography suggests evidence of cardiac involvement: the thickness of the interventricular septum and/or the posterior wall of the left ventricle is ≥ 12 mm.

Exclusion Criteria:

1. Amyloidosis is not caused by TTR protein, such as light chain amyloidosis;
2. There is meningeal transthyretin amyloidosis;
3. Allergic to any lipid nanoparticle (LNP) component or has previously received LNP and experienced treatment-related laboratory abnormalities or adverse events;
4. Use any of the following ATTR treatments within the prescribed time:

   * In the dose escalation stage of the first stage, the use history of Patisiran, Inotersen, and Vutrisiran is excluded;
   * In the dose expansion stage of the second stage, the following are excluded: Patisiran is used within 90 days before the administration of the investigational drug; Inotersen is used within 160 days before the administration of the investigational drug; Vutrisiran has a previous use history;
   * Tafamidis: used within 10 days before the administration of the investigational drug;
   * Diflunisal: used within 3 days before the administration of the investigational drug;
   * Doxycycline and/or taurodeoxycholic acid: used within 14 days before the administration of the investigational drug;
   * Previous use history of investigational gene editing drugs;
   * Other drugs for the treatment of ATTR: the last use is less than 30 days or 5 half-lives before the administration of the investigational drug, whichever is longer.
5. Unable or unwilling to supplement vitamin A during the trial;
6. History of multiple myeloma;
7. Ophthalmological examination results at the screening are consistent with vitamin A deficiency;
8. Abnormal thyroid function test with clinical significance judged by the investigator;
9. Known or suspected systemic infection (viral, parasitic or fungal infection) within 14 days before screening;
10. History of past hepatitis B virus, hepatitis C virus, acquired immunodeficiency syndrome or positive HBsAg, HCV-Ab, and HIV-Ab at the screening;
11. History of previous liver, heart or other organ transplantation or bone marrow transplantation or expected transplantation within 1 year (except for the history of corneal transplantation or planned corneal transplantation);
12. History of bleeding or coagulation disorders (such as cirrhosis, malignant hematological disease, antiphospholipid antibody syndrome);
13. History of acute thrombosis within 6 months before screening (such as acute myocardial infarction, acute cerebral infarction), or positive Leiden factor V and/or prothrombin gene test;
14. History of malignant tumor within 5 years before screening (except for basal cell carcinoma of the skin, radicalized squamous cell carcinoma of the skin, and carcinoma in situ of the cervix);
15. Planned invasive cardiovascular surgery during the trial (such as coronary artery stent/coronary artery bypass, pacemaker placement, etc.); those who have undergone cardiovascular invasive surgery within 90 days before screening or have been hospitalized due to heart failure;
16. History of alcohol abuse within 3 years before screening (definition of alcohol abuse: women drink ≥ 4 glasses/day or 8 glasses/week, men ≥ 5 glasses or 15 glasses/week, where 1 glass = 14g of pure alcohol);
17. Expected survival period is less than 1 year;
18. Other situations that the investigator deems inappropriate to enter this trial;

    For ATTR-PN only:
19. Other known diseases that cause motor or sensory neuropathy (such as diabetic neuropathy, neuropathy related to autoimmune diseases, etc.);
20. Diagnosed with type 1 diabetes or type 2 diabetes for ≥ 5 years;
21. NYHA cardiac function classification is grade III or IV within 90 days before screening;

    For ATTR-CM only:
22. NYHA cardiac function classification is grade IV within 90 days before screening;
23. PND score is grade IIIa, IIIb or IV at the screening;
24. Suffering from other cardiomyopathies not caused by TTR (such as hypertensive cardiomyopathy, valvular heart disease, cardiomyopathy caused by ischemic heart disease, etc.).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | through week 104
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Affiliated Hospital, School of Medicine, Zhejiang University, Hanzhou, Zhejiang